CLINICAL TRIAL: NCT03508713
Title: Long-term Prognosis and Quality of Life in Early Rheumatoid Arthritis Patients Treated by 2015 ACR Guideline (LELAND): a Multicenter Prospective Observational Study in Southern China
Brief Title: Long-term Prognosis and Quality of Life in Early Rheumatoid Arthritis Patients Treated by 2015 ACR Guideline (LELAND)
Acronym: LELAND
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Min Yang, Director, Head of Rheumatology, Principal Investigator, Clinical Professor, Nanfang Hospital, Southern Medical University
Other Study IDs: LC2016PY020
Record Dates: First submitted 2017-06-04; First posted 2018-04-26 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; prognosis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Biological Factors; Antirheumatic Agents; Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- early RA patients: patients must fulfill the 1987 ACR classification criteria for rheumatoid arthritis or 2010 Rheumatoid arthritis classification criteria of ACR/EULAR, and meet the condition that the course of disease was no more than 6 months. If enrolled, patients will be treated with disease modified antirheumatic drugs or biological agents.
  Interventions: Drug: disease modified antirheumatic drugs or biological agents

INTERVENTIONS:
Drug: disease modified antirheumatic drugs or biological agents — Enrolled patients will be treated according to the 2015 American College of Rheumatology Guideline for the Treatment of RA
  Other Names: DMARDs, MTX, biologics

SUMMARY:
To focus on the real world treat-to-target rate of early rheumatoid arthritis patients who will be treated according to the 2015 American College of Rheumatology Guideline for the Treatment of RA.

To explore the factors which influence the treat-to-target outcome.

DETAILED DESCRIPTION:
Resent study showed that rapid progression of cartilage and bone damage could happen on the early state of RA patients, so the clinicians should try the best to stop the trend, such as early diagnosis, early treatment and treat-to-target. But only half of the RA patients could reach low disease activity in the whole world and about 10% in China.

The investigators enroll early RA patients who are treated according to the 2015 American College of Rheumatology Guideline. The relevant data are collected and analyzed by the statistician including clinical data, imaging markers, blood samples and patient-reported outcomes every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years,
* be diagnosed with RA according to the 1987 or 2010 ACR criteria,
* in the course of the disease within 6 months,
* fill out questionnaires by oneself,
* fully understand the survey, agree to take part in the survey with signing the informed consent, and authority the researchers to expose and use his or her personal health information.

Exclusion Criteria:

* woman in pregnancy, lactation or plan to pregnant in the next 2 years,
* before enter this study, the patient joint any other RA clinical study in the past 24 weeks,
* according to the clinicians, one may not report his /or her life quality or the utilization of leading medical resources.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants entering this study are recruited from two hospital sites: Nanfang Hospital, Southern Medical University and Zhujiang Hospital, Southern Medical University.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-05-13 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients achieving treat to target | 2018-4-25 to 2022-7-1
  calculate the proportion of patients achieving treat to target according to the change of DAS28 score

SECONDARY OUTCOMES:
the change of Health Assessment Questionnaire Disability Index(HAQ-DI) | 2018-4-25 to 2022-7-1
  the change of Health Assessment Questionnaire Disability Index(HAQ-DI)
the change of The Work Productivity and Activity Impairment Questionnaire(WPAI) | 2018-4-25 to 2022-7-1
  the change of The Work Productivity and Activity Impairment Questionnaire(WPAI)
the change of European Quality of Life-5 Dimensions(EQ-5D) | 2018-4-25 to 2022-7-1
  the change of European Quality of Life-5 Dimensions(EQ-5D)
the change of Short Form 36 Health Survey Questionnaire(SF-36) | 2018-4-25 to 2022-7-1
  the change of Short Form 36 Health Survey Questionnaire(SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Min Yang, doctor, Principal Investigator — Nanfang Hospital, Southern Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao J, Zhan T, Zhu J, Fan M, Huang Q, Ren H, Wu J, Yu Q, Lin J, Ouyang Q, An S, Yang M. Long-term prognosis and quality of life in patients with early rheumatoid arthritis treated according to the 2015 ACR guideline (LELAND): protocol for a multicentre prospective observational study in Southern China. BMJ Open. 2018 Nov 15;8(11):e023798. doi: 10.1136/bmjopen-2018-023798. PMID 30446575